CLINICAL TRIAL: NCT02440113
Title: Post-operative CT Follow up Measurement After Nellix Endoprosthesis Implantation in Patients With Abdominal Aortic Aneurysms.
Brief Title: Post-operative CT Follow up After Nellix Endoprosthesis Implantation
Status: Completed | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Principal Investigator, Michel Reijnen, M.D., PhD, Rijnstate Hospital
Other Study IDs: WP-14-857
Record Dates: First submitted 2015-01-12; First posted 2015-05-12 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: Abdominal Aortic Aneurysm; Endovascular Aortic Repair; Nellix Endovascular Sealing
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Nellix: Patients with endovascular Nellix repair
  Interventions: Device: Nellix

INTERVENTIONS:
Device: Nellix — Nellix Implantation

SUMMARY:
Multicenter retrospective CT follow up after aortic aneurysm repair using Nellix Endoprosthesis.

DETAILED DESCRIPTION:
Rationale:

In patients with abdominal aortic aneurysms the Nellix Endoprosthesis aims to reduce post-operative complications and subsequent re-intervention rates. Using two stents covered with two polymer filled endobags used for sealing and excluding the aneurysm sac. Preliminary results show promising results in reducing these complications. The new endoprosthesis is not only different in treatment but also in follow up imaging. To date it is unknown how the stent, polymer filled endobags and aneurysm appear in CT imaging in short and long term follow up.

Objective:

To assess and describe the normal computed tomography (CT) appearance at 30 days and 1 year after implantation of the Nellix Endoprosthesis.

Study population:

Approximately a total of 100 patients who underwent endovascular aneurysm repair using Nellix endoprosthesis in three different hospitals. The population is comprised of approximately fifty patients from Rijnstate Ziekenhuis Arnhem and twenty-five each from St. Antonius Nieuwegein and St. Elisabeth Tilburg.

Design and methods:

The study is designed as a multicenter retrospective cohort. Using CT-scans from regular follow up dates (30 days and 1 year) imaging will be retrospectively assessed using medical imaging software. Main study endpoints are defined as followed:

1. Changes in the infrarenal neck morphology (below the renal arteries)
2. Changes in the thrombus in the aneurysm sac
3. Changes in the aneurysm wall and geometry
4. Changes in the cobalt-chromium stent and their lumen
5. Changes in the polymer-filled endobags Using anonymous patient data a database will be created an securely stored. Patient consent for study participation will be attained before accessing patient files.

Nature and extent of the burden and risk associated with participation, benefit and group relatedness:

The study will not bring an extra burden or risk for patients participating. Patients are encouraged to participate to improve insight for patients with the same disease and might improve health care in the future for this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent endovascular abdominal aneurysm repair using the Nellix endoprosthesis

Exclusion Criteria:

* No specific exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent Nellix endovascular aortic repair
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Changes in the infrarenal neck morphology (below the renal arteries) | 1 year
Changes in the thrombus in the aneurysm sac | 1 year
Changes in the aneurysm wall and geometry | 1 year
Changes in the cobalt-chromium stent and their lumen | 1 year
Changes in the polymer-filled endobags Using anonymous patient data a database will be created an securely stored. Patient consent for study participation will be attained before accessing patient files | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Michel Reijnen, MD, PhD, Principal Investigator — Rijnstate Hospital

IPD SHARING:
Plan to Share IPD: Undecided